CLINICAL TRIAL: NCT04912999
Title: The Inflammatory Bowel Diseases Remission Registry
Brief Title: Inflammatory Bowel Diseases Remission Registry
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0268-19-TLV
Record Dates: First submitted 2021-03-24; First posted 2021-06-03 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Crohn Disease; Ulcerative Colitis; Pouchitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Pouchitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The inflammatory bowel diseases (IBDs), ulcerative colitis (UC) and Crohn's disease (CD), are characterized by lifelong relapsing-remitting gastrointestinal inflammation, with symptoms of abdominal pain, diarrhea, and rectal bleeding during active disease. Medical therapy reduces intestinal inflammation and ameliorates symptoms. Clinical remission is defined when symptoms are resolved. In these periods, patients are able to perform daily activities more freely and lead a normal lifestyle. Biochemical remission (normalization of CRP and fecal Calprotectin) and endoscopic remission (no visual signs of inflammation of the mucosa in endoscopy) are the goals of IBD treatment.

Unfortunately, 30-40% of patients will relapse during 6 months from achieving remission. Risk factors for disease exacerbation are still unknown, and no guidelines exist as to the prevention of relapse and maintenance of remission in IBD patients.

In addition to the above, sleep disturbances and disturbances in the circadian rhythm can be a potential cause of flare-up. Sleep disorders cause changes in immune function, which later affect the course of the disease in IBD. This back affects the sleep pattern, so that a cycle is created, which may perpetuate the inflammation.

The interactions between sleep and inflammation are complex. An effective immune system affects sleep, and sleep disorders affect the functioning of the immune system. Furthermore, changes in the biological clock and sleep deprivation have been directly shown to worsen ulcerative colitis in laboratory animals. In people with sleep disorders, high levels of inflammation were found.

However, it is difficult to dissect the cause and effect for these associations, given their complex interactions.

Therefore we are planning to conduct a prospective study to assess variety of factors that might be associated with the activity of IBD.

DETAILED DESCRIPTION:
Prospectively follow IBD patients in remission (both clinical and biochemical) until disease exacerbation.

• Specific aims:

* To detect risk factors and early signs for disease exacerbation in IBD patients.
* To detect predictors of disease exacerbation from environmental and behavioral characteristics of patients, clinical and biochemical characteristics of the disease.
* To examine whether changes in circadian rhythm are associated with improvement in clinical and biological disease activity

Study design:

* A prospective cohort study. Eligible patients will be follow up for at least one year or until relapse time.
* Setting: prospectively collect clinical, behavioral, dietary and environmental data of IBD patients currently declared in an endoscopic remission according to the criteria in Israel. Data will be collected according to a uniform standardized protocol specifically adapted to the needs of the study. The team will include members of the IBD clinic at the Tel Aviv Medical Center, run by Dr. Nitsan Maharshak.

Study population:

Eligible IBD patients treated at the IBD clinic in the Tel Aviv Medical Center participating in the study, which have signed an informed consent form and answered to all the study inclusion criteria. Patients will be informed of the study by their treating physician, recruited and followed throughout the follow-up period by study co-ordinators.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as suffering from Crohn's disease (CD), Ulcerative colitis (UC) or Pouchitis for at least 2 months who are in clinical and biologic remission according to Steroid free clinical remission for greater or equal to 3 months according to the following activity index

  * Harvey Bradshaw index (HBI)<5 for CD patients
  * Simple Clinical Colitis activity index (SCCAI)≤2 for UC patients
  * Pouch disease activity index ≤6 / mPDAI ≤4 for Pouch patients

Also, patients will be included if they fullfull the following:

* Age 18-80 years
* Clinically stable patients, on constant medicinal regimen (mesalamine at least 4 weeks, or immunomodulators at least 12 weeks or biologics at least 12 weeks therapy, medical cannabis at least 2 weeks before inclusion to the study)

Exclusion Criteria:

* • Inability to sign an informed consent and complete the study protocol

  * Steroid therapy during the past 3 months
  * Antibiotic therapy during the past 2 weeks
  * Unstable or uncontrolled medical disorder, and sever systemic disease (other than IBD)
  * Participating in another clinical interventional trial
  * Stoma

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible IBD patients treated at the IBD clinic in the Tel Aviv Medical Center participating in the study, which have signed an informed consent form and answered to all the study inclusion criteria. Patients will be informed of the study by their treating physician, recruited and followed throughout the follow-up period by study co-ordinators.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Disease exacerbation for CD patients | follow up for at least one year or until relapse time or until 2 years of follow up
  Disease exacerbation by any of the following:
  * Increase in the specific clinical score:
    o Harvey Bradshaw index (HBI)≥5 for CD patients. HBI score ranges from 0 to 16 or more and the highest score depends on the number of liquid stools per day and indicates disease severity/activity
  * A change in disease activity requiring a change in medication, hospitalization, or a surgery.
  sample will be collected at baseline and follow up visits:
Disease exacerbation in UC patients | follow up for at least one year or until relapse time or until 2 years of follow up
  Disease exacerbation by any of the following:
  * Increase in the specific clinical score:
    o Simple Clinical Colitis activity index (SCCAI)>2 for UC patients. SCCAI score ranges from 0 to 19 and the highest score indicates disease severity/activity
  * A change in disease activity requiring a change in medication, hospitalization, or a surgery.
  sample will be collected at baseline and follow up visits:
Disease exacerbation in UC-Pouch patients | follow up for at least one year or until relapse time or until 2 years of follow up
  Disease exacerbation by any of the following:
  * Increase in the specific clinical score:
    o Pouch disease activity index (mPDAI) >4 for Pouch patients. mPDAI score ranges from 0 to 6 and the highest score indicates disease severity/activity
  * A change in disease activity requiring a change in medication, hospitalization, or a surgery.
  sample will be collected at baseline and follow up visits:

SECONDARY OUTCOMES:
nutritional factors as a risk of disease exacerbation | at baseline and follow up visits (until 2 years of follow up) or until relapse
  Questionnaires will be collected at baseline and follow up visits (dietary consumption)
  • Food frequency questionnaire, Processed foods questionnaire (PFQ), Lifestyle questionnaire
o Circadian rhythm as a risk factor for relapse | follow up for at least one year or until relapse time
  • Circadian rhythm questionnaire will be collected at baseline and foloow up visits
o Stress as a risk factor for relapse | follow up for at least one year or until relapse time
  • Promise questionnaire will be collected at baseline and follow up visits

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center; ,, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No